CLINICAL TRIAL: NCT00229892
Title: Small Incisions for Cardiac Surgery
Brief Title: Incisions for Cardiac Surgery
Status: Terminated | Type: Observational
Why Stopped: after 90 charts reviewed, insufficient data to support conclusion
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 04-120
Record Dates: First submitted 2005-09-13; First posted 2005-09-30 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2007-05

CONDITIONS: Cardiac Surgery; Cardiac Diseases
Keywords: pediatric health; cardiac; small incisions; operations; minimally invasive
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose is to evaluate the investigators' length of incisions based on patient weight, operative times, hospital lengths of stay, pain medicine requirements, complications and costs. These data will lead to a new minimally invasive standard of care without a reduction in outcomes.

DETAILED DESCRIPTION:
There is a trend in surgery, in general, toward minimal invasion. This includes the transition to laparoscopy/thoracoscopy from open procedures, as well as the reduction in incision size for open procedures. The goal of minimally invasive techniques is to reduce morbidity and length of hospital stay, with a consequent reduction in hospital cost.

There are few cardiac operations that are currently performed with minimally invasive techniques. One of these is the repair of an atrial septal defect, which can be performed though a small skin incision and partial rather than full sternotomy. Another is the ligation of a patent ductus arteriosus, which can be performed through a muscle-sparing thoracotomy rather than a full thoracotomy.

Both of these techniques minimize the scarring and the healing time required for post-operative recovery. We need to be confident that it has not affected our outcomes adversely. We need to evaluate our length of incisions based on patient weight, operative times, hospital lengths of stay, pain medicine requirements, complications and costs.

Hopefully, these data will lead to a new minimally invasive standard of care without a reduction in outcomes.

We will review charts before November 1, 2004 at Children's Healthcare of Atlanta.

ELIGIBILITY:
Inclusion Criteria:

* Children who have undergone cardiac surgery at Children's Healthcare of Atlanta
* Surgery before November 1, 2004

Exclusion Criteria;

those who do not fall under the above inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: children who have undergone cardiac surgery at Children's, Egleston, before 11.1.2004
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2005-02; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kogon, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States